CLINICAL TRIAL: NCT04348734
Title: Management of Parapneumonic Pleurisy Guided by an Early Pleural Ultrasound
Acronym: ECHOPP
Status: Completed | Type: Observational
Sponsor: Central Hospital Saint Quentin (Other Government)
Collaborators: Amiens University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-A00993-46
Record Dates: First submitted 2020-03-30; First posted 2020-04-16 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-03

CONDITIONS: Community-Acquired Infections
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pleural ultrasound — Patients will benefit from a daily pleural ultrasound for 96 hours, D1 being the day of hospitalization. The therapeutic course of action will depend on the presence or not, and on the type of pleural effusion according to a pre-established algorithm

SUMMARY:
Parapneumonic pleurisies are a frequent complication of pneumopathies, but therapeutic management is poorly codified. Only the indication of thoracic drainage has benefited from expert recommendations. However, we find in the literature the major importance of early management of infectious pleurisy in order to minimize the sequelae. Pleural ultrasound, sensitive and specific in this pathology could bring us a real interest in terms of diagnostic speed and therefore of care. This study therefore seeks to show that pleural ultrasound can have a major interest in improving the management of patients with parapneumonic pleurisy, by reducing the number of medical treatment failures.

DETAILED DESCRIPTION:
This is a prospective, multicentre, non-randomized study evaluating routine care, which includes all patients hospitalized in the departments participating in the study, for pneumonia with or without pleurisy. Patients benefiting from a daily pleural ultrasound for 96 hours, D1 being the day of hospitalization. The therapeutic course of action will depend on the presence or not, and on the type of pleural effusion according to a pre-established algorithm. In case of pleural effusion of type 1, the type of treatment will be left to the appreciation of the clinician (puncture or drainage), in case of pleural effusion of type 2, 3 or 4 the patient benefited from pleural drainage.

Patients included in the study will benefit from a pleural ultrasound on the day of their hospitalization, up to 96 hours after treatment. Ultrasound will then allow us to look for the presence of pleural effusion. In the event of effusion corresponding to a parapneumonic effusion or purulent pleurisy, the conduct to be followed will be defined according to the ultrasound type of effusion. Types 1 will benefit from an evacuating pleural puncture or drainage, depending on the clinician's judgment. Types 2, 3, and 4 will benefit from weeping drainage.

the target population: adult patients, hospitalized for pneumonia or confirmed pleurisy, by imaging and exploratory pleural puncture in the departments participating in the study over the period concerned The main outcome measure is the failure of medical treatment, defined as the need to resort to surgery, with or without peeling, or death secondary to pleurisy. The secondary endpoint is the presence of radiological sequelae at 3 months and 6 months defined by a retraction of the hemithorax concerned with pachypleuritis or an ascent of the diaphragmatic dome or the persistence of pleurisy

ELIGIBILITY:
Inclusion Criteria:

* adult patients, hospitalized for pneumonia or confirmed pleurisy, by imaging and exploratory pleural puncture.
* Patients affiliated to social security

Exclusion Criteria:

* patients with transudative pleurisy,
* patients with exudative pleurisy in the context of pulmonary neoplasia or tuberculosis,
* patients with pneumonectomy compartment infections,
* Patient under guardianship or curatorship,
* Subjects under 18 years of age,
* Pregnant women,
* patients in emergency situations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for pneumonia
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
interet de l'échographie pleurale dans les pleurésies parapneumoniques | 1 year
  Evaluate the failure of medical treatment, defined as the need to resort to surgery, or death secondary to pleuris

SECONDARY OUTCOMES:
presence radiological sequelae a pleural effusion at 3 months | 3 months
  the presence of radiological sequelae at 3 months defined by a retraction of the hemithorax concerned with pachypleuritis or an ascent of the diaphragmatic dome or the persistence of a pleural effusion
presence radiological sequelae a pleural effusion at 6 months | 6 months
  the presence of radiological sequelae at 6 months defined by a retraction of the hemithorax concerned with pachypleuritis or an ascent of the diaphragmatic dome or the persistence of a pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: DOUADI Dr Youcef, ch, Principal Investigator — CH SAINT-QUENTIN
Locations (4):
- France (4):
  - Chu Amiens, Amiens
  - CH Pontoise, Cergy-Pontoise
  - CH Creteil, Créteil
  - Saint-Quentin Hospital, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No
the data will be collected on an electronic Ecrf, a single extraction is planned by the protocol, all the collected data will be analyzed centrally by the study cordernator,no data sharing is planned in the study

REFERENCES:
- [Result] Light RW. Pleural diseases. Curr Opin Pulm Med. 2003 Jul;9(4):251-3. doi: 10.1097/00063198-200307000-00001. No abstract available. PMID 12806235
- [Result] Miserocchi G. Physiology and pathophysiology of pleural fluid turnover. Eur Respir J. 1997 Jan;10(1):219-25. doi: 10.1183/09031936.97.10010219. PMID 9032518
- [Result] Davies CW, Gleeson FV, Davies RJ; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of pleural infection. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii18-28. doi: 10.1136/thorax.58.suppl_2.ii18. No abstract available. PMID 12728147
- [Result] Hamm H, Light RW. Parapneumonic effusion and empyema. Eur Respir J. 1997 May;10(5):1150-6. doi: 10.1183/09031936.97.10051150. PMID 9163661
- [Result] LeMense GP, Strange C, Sahn SA. Empyema thoracis. Therapeutic management and outcome. Chest. 1995 Jun;107(6):1532-7. doi: 10.1378/chest.107.6.1532. PMID 7781342
- [Result] Bober K, Swietlinski J. Diagnostic utility of ultrasonography for respiratory distress syndrome in neonates. Med Sci Monit. 2006 Oct;12(10):CR440-6. Epub 2006 Sep 25. PMID 17006405
- [Result] Soldati G, Sher S. Bedside lung ultrasound in critical care practice. Minerva Anestesiol. 2009 Sep;75(9):509-17. PMID 19644435
- [Result] Ramnath RR, Heller RM, Ben-Ami T, Miller MA, Campbell P, Neblett WW 3rd, Holcomb GW, Hernanz-Schulman M. Implications of early sonographic evaluation of parapneumonic effusions in children with pneumonia. Pediatrics. 1998 Jan;101(1 Pt 1):68-71. doi: 10.1542/peds.101.1.68. PMID 9417153
- [Result] Xirouchaki N, Magkanas E, Vaporidi K, Kondili E, Plataki M, Patrianakos A, Akoumianaki E, Georgopoulos D. Lung ultrasound in critically ill patients: comparison with bedside chest radiography. Intensive Care Med. 2011 Sep;37(9):1488-93. doi: 10.1007/s00134-011-2317-y. Epub 2011 Aug 2. PMID 21809107
- [Result] Tokuda Y, Matsushima D, Stein GH, Miyagi S. Intrapleural fibrinolytic agents for empyema and complicated parapneumonic effusions: a meta-analysis. Chest. 2006 Mar;129(3):783-90. doi: 10.1378/chest.129.3.783. PMID 16537882
- [Result] Stavas J, vanSonnenberg E, Casola G, Wittich GR. Percutaneous drainage of infected and noninfected thoracic fluid collections. J Thorac Imaging. 1987 Jul;2(3):80-7. doi: 10.1097/00005382-198707000-00011. PMID 3302292
- [Result] Sahn SA. Management of complicated parapneumonic effusions. Am Rev Respir Dis. 1993 Sep;148(3):813-17. doi: 10.1164/ajrccm/148.3.813. No abstract available. PMID 8368654
- [Result] Taryle DA, Potts DE, Sahn SA. The incidence and clinical correlates of parapneumonic effusions in pneumococcal pneumonia. Chest. 1978 Aug;74(2):170-3. doi: 10.1378/chest.74.2.170. No abstract available. PMID 679746
- [Result] Pothula V, Krellenstein DJ. Early aggressive surgical management of parapneumonic empyemas. Chest. 1994 Mar;105(3):832-6. doi: 10.1378/chest.105.3.832. PMID 8131548
- [Result] Saito T, Kobayashi H, Kitamura S. Ultrasonographic approach to diagnosing chest wall tumors. Chest. 1988 Dec;94(6):1271-5. doi: 10.1378/chest.94.6.1271. PMID 3056662
- [Result] Lichtenstein DA. BLUE-protocol and FALLS-protocol: two applications of lung ultrasound in the critically ill. Chest. 2015 Jun;147(6):1659-1670. doi: 10.1378/chest.14-1313. PMID 26033127
- [Result] Lichtenstein DA, Menu Y. A bedside ultrasound sign ruling out pneumothorax in the critically ill. Lung sliding. Chest. 1995 Nov;108(5):1345-8. doi: 10.1378/chest.108.5.1345. PMID 7587439